CLINICAL TRIAL: NCT05028595
Title: Evaluation of Hepatic Affection in Hemodialysis Patients With Iron Overload in Assiut University Hospital
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa M.Abokresha, principle investigator, Assiut University
Other Study IDs: Hepatic MRI
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Hepatic Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim of the work

1. Assessment of hepatic affection in patients with ESRD (end stage renal disease) on regular dialysis with iron indices suggesting iron overload.
2. Comparison between HCV -negative HD patients with high and normal TSAT as regard liver iron concentration(LIC) and degree of fibrosis.

DETAILED DESCRIPTION:
Anemia is a common complication in patients with chronic kidney disease (CKD) . The main cause of anemia is the inadequate production of erythropoietin. Iron deficiency is another common cause of anemia in these patients . Inflammation is another hallmark of CKD that may lead to a "functional" iron deficient anemia .

The first treatment used to correct anemia in CKD patients was blood transfusion. However, the risk of transfusion reaction, transmission of infectious agents and iron overload triggered the search for a better treatment of anemia .

Nowadays, the gold standard treatment for anemia in CKD patients is the administration of erythropoiesis stimulating agents (ESAs), associated with iron supplementation . Although the majority of the patients respond to ESA therapy, about 10% of CKD patients are hypo-responsive . One of the causes for hypo-responsiveness to ESAs is iron deficiency, either absolute or functional . A ferritin value lower than 30 ng/mL in men or lower than 15 ng/mL in women are consistent with absolute iron deficiency ; a serum ferritin concentration higher than 300 ng/mL, along with anemia, indicates a functional iron deficiency, as it usually occurs in CKD patients .

The "Clinical Practice Guideline for Anemia in Chronic Kidney Disease" from KDIGO stated that CKD patients with anemia should first start iron therapy rather than ESAs .

The Dialysis Outcomes and Practice Patterns Study (DOPPS) showed that the number of HD patients with IV iron supplementation increased in most countries and the doses prescribed to these patients also increased in the past 10-15 years.

The liver is the main site of iron storage, and the liver iron concentration (LIC) is closely correlated with total body iron stores in patients with secondary forms of hemosiderosis such as thalassemia major, sickle cell disease, and genetic hemochromatosis . Non-invasive techniques for estimating liver iron stores have been developed to avoid liver biopsy, including the superconducting quantum interference device (SQUID), quantitative computed tomography, and MRI .

More than one study show that 84% of the HD patients had hepatic iron overload, and in 30% of them iron overload was severe; moreover, iron liver content correlated with infused iron .

In spite of the widespread use of IV iron supplementation in HD patients, the safest dosing strategy is still poorly clarified, as well as its relation with serum ferritin levels, iron overload and mortality risk.

ELIGIBILITY:
Inclusion Criteria:

* Eighty patients with end-stage kidney disease (ESKD) on regular hemodialysis for more than two years were enrolled in the study with normal serum ferritin level at the start of dialysis

Exclusion Criteria:

* Patients with one or more of the following conditions were excluded; non-dialysis-dependent chronic kidney disease patients (NDD-CKD), iron deficiency anaemia (diagnosed based on iron studies included serum iron, ferritin and total iron binding capacity), other causes of hemochromatosis such as genetic type, or hemochromatosis secondary to hemolytic anemia, hepatitis B virus infection, and human immunodeficiency virus infection. Moreover, patients with additional causes of liver disease, including non-alcoholic fatty liver disease, primary sclerosing cholangitis, primary biliary cholangitis, etc. were excluded.

Other exclusion criteria included active malignancy, heart failure, use of immunosuppressive drugs, previous liver transplantation, and patients who are below 18 year of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PT with ESRD on regular haemodialysis
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Assessment of hepatic affection in patients with ESRD (end stage renal disease) on regular dialysis with iron indices suggesting iron overload. | Baseline
  MRI for abdomen was done .patient on supine position and multiple cuts were taken

SECONDARY OUTCOMES:
Comparison between HCV -negative HD patients with high and normal TSAT as regard liver iron concentration(LIC) and degree of fibrosis. | Baseline
  Assesment of degree of hepatic fibrosis by fibroscan machine ,Patients on supine position and sonar probe placed between ribs9-11 to asses degree of fibrosis

CONTACTS AND LOCATIONS:
Locations (1):
- Marwa Abokresha, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stauffer ME, Fan T. Prevalence of anemia in chronic kidney disease in the United States. PLoS One. 2014 Jan 2;9(1):e84943. doi: 10.1371/journal.pone.0084943. eCollection 2014. PMID 24392162
- [Background] Ribeiro S, Belo L, Reis F, Santos-Silva A. Iron therapy in chronic kidney disease: Recent changes, benefits and risks. Blood Rev. 2016 Jan;30(1):65-72. doi: 10.1016/j.blre.2015.07.006. Epub 2015 Aug 18. PMID 26342303
- [Background] Nangaku M, Eckardt KU. Pathogenesis of renal anemia. Semin Nephrol. 2006 Jul;26(4):261-8. doi: 10.1016/j.semnephrol.2006.06.001. PMID 16949463
- [Background] Costa E, Lima M, Alves JM, Rocha S, Rocha-Pereira P, Castro E, Miranda V, do SF, Loureiro A, Quintanilha A, Belo L, Santos-Silva A. Inflammation, T-cell phenotype, and inflammatory cytokines in chronic kidney disease patients under hemodialysis and its relationship to resistance to recombinant human erythropoietin therapy. J Clin Immunol. 2008 May;28(3):268-75. doi: 10.1007/s10875-007-9168-x. PMID 18205031
- [Background] do Sameiro-Faria M, Ribeiro S, Costa E, Mendonca D, Teixeira L, Rocha-Pereira P, Fernandes J, Nascimento H, Kohlova M, Reis F, Amado L, Bronze-da-Rocha E, Miranda V, Quintanilha A, Belo L, Santos-Silva A. Risk factors for mortality in hemodialysis patients: two-year follow-up study. Dis Markers. 2013;35(6):791-8. doi: 10.1155/2013/518945. Epub 2013 Nov 24. PMID 24347799
- [Background] Lukaszyk E, Lukaszyk M, Koc-Zorawska E, Tobolczyk J, Bodzenta-Lukaszyk A, Malyszko J. Iron Status and Inflammation in Early Stages of Chronic Kidney Disease. Kidney Blood Press Res. 2015;40(4):366-73. doi: 10.1159/000368512. Epub 2015 Jun 20. PMID 26160488
- [Background] Ibrahim HN, Ishani A, Guo H, Gilbertson DT. Blood transfusion use in non-dialysis-dependent chronic kidney disease patients aged 65 years and older. Nephrol Dial Transplant. 2009 Oct;24(10):3138-43. doi: 10.1093/ndt/gfp213. Epub 2009 May 18. PMID 19451656
- [Background] Drueke TB, Parfrey PS. Summary of the KDIGO guideline on anemia and comment: reading between the (guide)line(s). Kidney Int. 2012 Nov;82(9):952-60. doi: 10.1038/ki.2012.270. Epub 2012 Aug 1. PMID 22854645
- [Background] Kuwahara M, Mandai S, Kasagi Y, Kusaka K, Tanaka T, Shikuma S, Akita W. Responsiveness to erythropoiesis-stimulating agents and renal survival in patients with chronic kidney disease. Clin Exp Nephrol. 2015 Aug;19(4):598-605. doi: 10.1007/s10157-014-1023-9. Epub 2014 Sep 3. PMID 25183365
- [Background] National Kidney Foundation. K/DOQI clinical practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Am J Kidney Dis. 2002 Feb;39(2 Suppl 1):S1-266. No abstract available. PMID 11904577